CLINICAL TRIAL: NCT05692388
Title: Mixed Methods Study of Health-Related Social Needs in African American Adults With Chronic Kidney Disease and Type 2 Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Mukoso N. Ozieh, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00043301; 1K23MD016448-01A1 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Nephropathy Type 2 - Uncontrolled; Diabetes Mellitus, Type 2; Chronic Kidney Diseases
Keywords: Social risk factors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aim 1: Qualitative Aim
  Interventions: Other: Patient and Community Stakeholder Interviews
- Aim 2: Quantitative Aim
  Interventions: Other: Cross-sectional Study Participants
- Aim 3: Integrative Aim
  Interventions: Other: Focus Groups and Intervention Mapping

INTERVENTIONS:
Other: Patient and Community Stakeholder Interviews — Thirty in-depth face-to-face patient interviews, and ten in-depth structured stakeholder interviews will be conducted to explore and identify facilitators and barriers to self-care in African American adults with DKD experiencing HRSN.
  Groups: Aim 1
Other: Cross-sectional Study Participants — Three hundred African American adults with DKD experiencing HRSN will be recruited to participate in a cross-sectional study. All participants will complete a one-time survey, and blood samples and blood pressure readings will be obtained to assess clinical outcomes.
  Groups: Aim 2
Other: Focus Groups and Intervention Mapping — A subsample of patient interview/cross-sectional study participants will be invited back to participate in four focus groups (five participants/group) to review components of the intervention, give feedback on appropriateness, feasibility, acceptability, and likelihood of having an impact based on their lived experiences.
  Groups: Aim 3

SUMMARY:
The overarching goal of this study is to understand facilitators and barriers to self-care, develop and refine a culturally tailored intervention to improve clinical outcomes, quality of life (QOL), and self-care behaviors in African American adults with diabetic kidney disease (DKD) experiencing health-related social needs (HRSN).

DETAILED DESCRIPTION:
Health-related social needs (HRSN) including loss of employment, housing instability, food insecurity, transportation needs, utility needs, interpersonal safety, and financial strain impacts the complex self-management of DKD such as self-monitoring and behavior modification. This study utilizes a convergent parallel mixed methods study design to understand facilitators and barriers to care and develop a culturally tailored intervention to improve clinical outcomes, quality of life, and self-care behaviors in African American adults with DKD experiencing HRSN.

Aim 1 (Qualitative): Identify facilitators and barriers to care in African American adults with DKD experiencing HRSN using in-depth patient and stakeholder interviews.

Aim 2 (Quantitative): Examine the effect of increasing burden of HRSN on clinical outcomes (hemoglobin A1c, blood pressure, lipids), quality of life, and self-care behaviors (diet, exercise, and medication adherence) in a sample of 300 African American adults with DKD experiencing HRSN.

Aim 3 (Integrative): Integrate findings from Aims 1 and 2 and develop a culturally tailored intervention to improve clinical outcomes, quality of life, and self-care behaviors in African American adults with DKD experiencing HRSN.

ELIGIBILITY:
Inclusion Criteria:

1. self- report as AA/Black
2. age ≥18
3. screen positive for 1 or more adversities using the Centers for Medicare and Medicaid Services Accountable Health Communities Health-Related Social Needs Screening tool
4. self-reported type 2 diabetes and self-report or screen positive for chronic kidney disease (CKD)
5. able to communicate in English.

Exclusion Criteria:

1. cognitive impairment at screening visit
2. active psychosis
3. active alcohol or drug abuse/dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include African American adults with diagnosed diabetic kidney and reporting multiple social risk factors.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | Baseline
  Blood pressure readings will be obtained using automated BP monitors
Hemoglobin A1c (HbA1c) | Baseline
  Blood sample will be drawn by a trained phlebotomist and sent to the laboratory for HbA1c.
LDL cholesterol | Baseline
  Blood sample will be drawn by a trained phlebotomist and sent to the laboratory for LDL cholesterol.
Quality of Life (QOL) | Baseline
  Quality of Life will be assessed using SF-12, a valid and reliable instrument to measure functional status. This 12-item scale is a valid and reliable instrument of functional status and provides a summary physical health-related quality of life (PCS) and mental health-related quality of life (MCS). Scores for each of the PCS and MCS range from 0 to 100, with higher scores indicating better physical and mental health-related quality of life, respectively.
Self-Care Behavior | Baseline
  Self-Care Behavior will be assessed with the Summary of Diabetes Self-Care Activities scale. This is an 11-item self-reported questionnaire including items assessing diet, exercise, blood glucose test, foot care, and smoking status. Higher scores indicate more engagement in self-care behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Mukoso N Ozieh, MD, MSCR, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States